CLINICAL TRIAL: NCT01343784
Title: Assessment of Voiding After Sling (AVAS): A Randomized Trial of Two Methods of Post-operative Catheter Management After Midurethral Sling for Female Stress Urinary Incontinence
Brief Title: Assessment of Voiding After Sling
Acronym: AVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: IRB 11-082
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Post-operative Voiding
Keywords: Voiding trial; sling; post-operative assessment; urinary retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Voiding Trial (Active Comparator): Subjects in this group will undergo backfill-assisted voiding trial that involves infusing 300ml of fluid in the bladder, removing the catheter and allowing the patient to void. All subjects will be asked to use visual analog scale (VAS) to assess their force of stream (FOS) and the voided amount as well as post-void residual (PVR) (measured by the bladder ultrasound) will be measured and recorded. Subjects will be discharged without a catheter if the voided amount is more than 200ml, or 2/3rds of the infused volume (300ml).
  Interventions: Other: Urinary voiding assessment after midurethral sling
- Force of Stream Voiding Trial (Experimental): Subjects in this group will undergo backfill-assisted voiding trial that involves infusing 300ml of fluid in the bladder, removing the catheter and allowing the patient to void. All subjects will be asked to use visual analog scale (VAS) to assess their force of stream (FOS) and the voided amount as well as post-void residual (PVR) (measured by the bladder ultrasound) will be measured and recorded. Subjects in the FOS group will be discharged home without a catheter if they are able to void any amount and report an FOS of at least 50% their typical FOS based on a visual analog scale
  Interventions: Other: Urinary voiding assessment after midurethral sling

INTERVENTIONS:
Other: Urinary voiding assessment after midurethral sling — Both groups will undergo voiding trial in the similar manner. The decision to discharge based on an objective measure (voided amount) versus based on the subjective measure (force of stream self assessment).

SUMMARY:
The purpose of this study is to compare the incidence of catheterization from discharge to 6 weeks postoperatively when using two methods of post-operative voiding evaluation after a mid-urethral sling procedure. The investigators' results may lead to a decreased use of indwelling catheters and their associated morbidity after outpatient sling surgery.

DETAILED DESCRIPTION:
Minimally invasive slings have demonstrated similar efficacy to earlier abdominal anti-incontinence procedures, but offer the benefit of shorter operating times, less voiding dysfunction, lower morbidity and are usually done as an outpatient procedure. Despite the advantages, about 35% of patients are discharged home with indwelling catheters. Indwelling catheters are bothersome for patients, costly to the healthcare system and are a source of significant morbidity. The challenge for pelvic surgeons performing anti-incontinence procedures is avoiding postoperative urinary retention while minimizing the use of catheters and their associated risks. A commonly described backfill-assisted voiding trial is used as a means of evaluating bladder function postoperatively. This method uses a low post-void residual as a specific criterion for discharge without a catheter. However, the validity of this method has never been critically evaluated. Our recent observational study suggests that patients may be safely discharged without a catheter after a midurethral sling procedure based on their subjective assessment of the force of stream. Our proposed study expands on this pilot data using a randomized trial to evaluate two methods of post-operative voiding evaluation. The results may lead to a decreased use of indwelling catheters and their associated morbidity after outpatient sling surgery.

ELIGIBILITY:
Enrollment:

All patients,18-81 year old, undergoing an outpatient midurethral sling surgery will be screened for participation in the study at the preoperative visit.

Exclusion:

1. Women undergoing concomitant urinary tract or pelvic reconstructive procedures
2. Women with pelvic organ prolapse beyond the hymen
3. Women who have undergone a different or same procedure for urinary incontinence in the past
4. Women with neurological conditions, such as multiple sclerosis, spinal cord injury/pathology
5. Cases complicated by a cystotomy or other complication necessitating postoperative catheterization
6. Non-English speakers

Ages: 18 Years to 81 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Total Catheterization Rate | Surgery to 6-weeks post-operatively
  The incidence of postoperative catheterization (total catheterization) at any point from discharge after surgery to 6 weeks postoperatively.
  The incidence of being discharged with an indwelling catheter will be gathered from PACU records. The information regarding catheterization after that point will be captured via the electronic medical records or patient questionnaires (at 2 days, 1 week, and 6 week follow-up).

SECONDARY OUTCOMES:
Subjective assessment of Force of Stream (FOS). | 30 minutes to 2 hours in recovery room
  Using VAS, the subject compares the post-operative FOS with the pre-operative FOS on a scale of 0-120% given the pre-operative FOS is 100%.
Number of return visits to the office or to the emergency room | 6 weeks
  This information will be captured via the EMR or the patient questionnaires, at 2-days, 1-week and 6-weeks folow-up.
Cumulative number of days of catheterization | 6 weeks
  Calculated from EMR at the 6-weeks post-operative visit.
Incidence of catheter acquired urinary tract infection (CAUTI) | 6 weeks
  UTI is defined according to the CDC as a positive culture >10^5 CFU/ml with no more than 2 species of microorganisms in the patient's endorsing 1 or more UTI symptoms.
Time to discharge from PACU | 30 minutes to 2 hours in recovery room
  Collected from EMR.
Effectiveness of the sling procedure | 6 weeks
  Incontinence severity index will be collected at enrollment and at 6 weeks post surgery. The score will be compared to determine if the procedure was effective at treating incontinence.
Postoperative pain | 6 weeks
  Pain scale will be administered at 2-days, 1-week and 6-weeks follow-up.
Patient's expectation of postoperative recovery | Assessed at enrollment, average 10 minutes
  Information will be collected via short survey at enrollment. The subject will be asked to assign a level of importance to post-operative factors such as pain control, prolonged catheterization, daily activities and ability to return to work.
Daily function postoperatively as well as satisfaction with the surgery | 6 weeks
  Information will be gathered from questionnaires at 2-days, 1-week and 6-weeks follow-up. Modified validated questionnaire will be used (McCarthy et al).

CONTACTS AND LOCATIONS:
Overall Officials: John Eric Jelovsek, MD, Principal Investigator — The Cleveland Clinic; Matthew Barber, MD, MHS, Study Director — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Beachwood, Beachwood, Ohio
  - Cleveland Clinic Hillcrest Hospital, Mayfield Heights, Ohio

REFERENCES:
- [Derived] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837